CLINICAL TRIAL: NCT02194673
Title: Acute Effects of Natural and Interesterified Fats-formulated Margarine on Lipemic and Insulinemic Response
Brief Title: Acute Effects of Natural and Interesterified Fats-margarine on Lipemic and Insulinemic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malaysia Palm Oil Board (Other Government)
Collaborators: IMU University, Malaysia (Other); Universiti Putra Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: AH 00112
Record Dates: First submitted 2014-06-25; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Trans free palm margarine (Experimental): One high fat muffin will be serves together with a glass of low fat milk shake.
  Interventions: Other: Trans free palm margarine; Other: Interesterified Palm based margarine; Other: IE Soybean oil-based margarine
- Interesterified palm based margarine (Experimental): One high fat muffin will be serves together with a glass of low fat milk shake.
  Interventions: Other: Trans free palm margarine; Other: Interesterified Palm based margarine; Other: IE Soybean oil-based margarine
- IE soybean oil-based margarine (Experimental): One high fat muffin will be serves together with a glass of low fat milk shake.
  Interventions: Other: Trans free palm margarine; Other: Interesterified Palm based margarine; Other: IE Soybean oil-based margarine

INTERVENTIONS:
Other: Trans free palm margarine — A randomised, double-blind crossover (3 × 3 arms) orthogonal Latin-square design was used and conducted on 10 males and 10 females adults.
Other: Interesterified Palm based margarine — A randomised, double-blind crossover (3 × 3 arms) orthogonal Latin-square design was used and conducted on 10 males and 10 females adults.
Other: IE Soybean oil-based margarine — A randomised, double-blind crossover (3 × 3 arms) orthogonal Latin-square design was used and conducted on 10 males and 10 females adults.

SUMMARY:
Interesterified (IE) fat blends will respond differently in terms of postprandial lipemia and insulinemic responses compare to a trans free palm margarine (TFPM).

DETAILED DESCRIPTION:
The objective of this study was to investigate whether IE-fat blends behave differently on postprandial serum lipid, insulin, C-peptide and glucose concentration compare to TFPM. A randomised, double-blind crossover (3 × 3 arms) orthogonal Latin-square design was used and conducted on 10 males and 10 females adults. During postprandial challenge day, each subject received an a test muffin incorporated with test margarine. Blood samples were collected at half-hourly intervals until 4 hr by using cannulation technique.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18.5 and 24.9
* <130mmHg for systolic pressure and <80 mmHg for diastolic pressure
* Blood glucose level in the range of 3.9 to 5.5 mmol/L
* Total cholesterol less than 5.17 mmol/L
* No use of tobacco and no consumption of alcohol.

Exclusion Criteria:

* Suffer from chronic disease
* Metabolic syndrome
* Consuming any medical prescriptions
* People with blood clotting problem
* Women who are pregnant
* Hypertensive person

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in serum triglycerides level of subjects as a measure of postprandial triglycerides response | Baseline, 4 hours

SECONDARY OUTCOMES:
Change in the level of plasma insulin, c-peptide and serum glucose as a measure of postprandial insulinemic response | Baseline, 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Voon Phooi Tee, Ph.D, Principal Investigator — Malaysia Palm Oil Board
Locations (1):
- MalaysiaPOB, Kajang, Selangor, Malaysia